CLINICAL TRIAL: NCT04574505
Title: Evaluation of the Effect of a Food Supplementation With Eufortyn Colesterolo Plus on the Modulation of LDL Cholesterolemia in Subjects Affected by Polygenic Hypercholesterolemia: a Two-arm Double-blind, Placebo- Controlled, Randomized, Clinical Trial.
Brief Title: Food Supplementation With Eufortyn Colesterolo Plus for LDL Modulation in Subjects With Polygenic Hypercholesterolemia
Acronym: ANEMONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: SCHARPER Spa (Unknown)
Responsible Party: Principal Investigator, Arrigo F.G. Cicero, Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCH 01/2020
Record Dates: First submitted 2020-09-14; First posted 2020-10-05 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: This is a two-arm randomized, placebo-controlled, double-blind, monocentric parallel-groups clinical study conducted in Italy.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NUT (Experimental): 1 tablet of Eufortyn Colesterolo Plus per day + standard diet for 8 weeks
  Interventions: Dietary Supplement: Eufortyn Colesterolo Plus
- Placebo (Placebo Comparator): 1 tablet of Placebo per day + standard diet for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Eufortyn Colesterolo Plus — Food supplement combination containing bergamot (Vazguard®) phytosomal polyphenolic fraction associated with standardized artichoke extract (Pycrinil®, Cynara Cardunculus L) and Cynara scolimus, associated with high coenzyme Q10 bioavailability(Q10 phytosome® Ubiqsome) and zinc.
  Arms: NUT
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a two-arm randomized, placebo-controlled, double-blind, monocentric parallel-groups clinical study conducted in Italy.

The objective of this study is to evaluate the effect of dietary supplementation of a combined supplement containing bergamot (Vazguard®) phytosomal polyphenolic fraction associated with standardized artichoke extract (Pycrinil®, Cynara cardunculus) and Cynara scolimus, associated with high coenzyme Q10 bioavailability (Q10 phytosome® Ubiqsome) and zinc, on the glycometabolic structure of subjects with suboptimal levels of LDL cholesterolemia compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects agree to participate in the study and having dated and signed the informed consent form.
* Subjects who have the capability to communicate, to make themselves understood, and to comply with the study's requirements.
* Male or female aged ≥ 18 years and ≤ 70 years old.
* LDL-Cholesterol plasma levels >115 mg/dL and < 190 mg/dL.
* TG<400 mg/dL.
* Subjects who, according to the SCORE charts, have a low or moderate cardiovascular risk (defined as a total cardiovascular risk < 5%) and for whom, according to ESC/EAS guidelines 2019, the intervention strategy does not require a pharmacological lipid lowering intervention.

Exclusion Criteria:

* Subjects already affected by cardiovascular diseases (secondary prevention) or with estimated 10 years cardiovascular disease risk> 5%;
* Obesity (BMI>30 kg/m2) or diabetes mellitus;
* Assumption of lipid lowering drugs or food supplements, or drugs potentially affecting the lipid metabolism;
* Antihypertensive treatment not stabilized since at least 3 months;
* Anticoagulants therapy
* Uncontrolled hypertension (systolic blood pressure> 190 mmHg or diastolic arterial pressure> 100 mmHg);
* Known current thyroid, gastrointestinal or hepatobiliary diseases;
* Any medical or surgical condition that would limit the patient adhesion to the study protocol;
* Abuse of alcohol or drugs (current or previous);
* History of malignant neoplasia in the 5 years prior to enrolment in the study;
* History or clinical evidence of inflammatory disease such as severe arthritis, systemic lupus erythematosus or chronic inflammatory diseases or current therapy with immunosuppressive agents or long-term glucocorticoids;
* History or clinical evidence of any significant concomitant disease that could compromise the safety of the subject or the possibility of completing the study;
* Known previous intolerance to one component of the tested nutraceuticals
* Women in fertile age not using consolidated contraceptive methods
* Pregnancy and Breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
The primary objective is to compare the effect on LDL-cholesterol after 8 weeks of treatment with a combined food supplement with placebo (standard diet only). | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arrigo Cicero, MD, Principal Investigator — University of Bologna
Locations (1):
- AOU Policlinico S.Orsola-Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fogacci F, Rizzoli E, Giovannini M, Bove M, D'Addato S, Borghi C, Cicero AFG. Effect of Dietary Supplementation with Eufortyn(R) Colesterolo Plus on Serum Lipids, Endothelial Reactivity, Indexes of Non-Alcoholic Fatty Liver Disease and Systemic Inflammation in Healthy Subjects with Polygenic Hypercholesterolemia: The ANEMONE Study. Nutrients. 2022 May 18;14(10):2099. doi: 10.3390/nu14102099. PMID 35631240